CLINICAL TRIAL: NCT05254730
Title: Using Micro-filaments to Detect "fast Ripples" and Improve the Identification of the Epileptogenic Zone
Acronym: NeuroSeizure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adrien Peyrache (Other)
Responsible Party: Sponsor-Investigator, Adrien Peyrache, Associate Professor, McGill University
Organization: McGill University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-5000
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy, Refractory
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- micro-macroelectrodes (Experimental): Patients will be implanted with usually the novel intracerebral micro-macroelectrodes (instead of the regular clinical macroelectrodes). The primary and secondary outcomes will then be assessed.
  Interventions: Device: macro-micro tetrodes for intracranial recording

INTERVENTIONS:
Device: macro-micro tetrodes for intracranial recording — novel design of tetrode micro electrodes within the standard macro intracranial electrodes used clinically for identification of the epileptogenic zone

SUMMARY:
record fast ripples with novel intracranial electrodes with micro-tetrodes to improve the identification of epileptogenic zone (EZ) and investigate the neuronal circuits underlying brain dynamics associated with epilepsy

DETAILED DESCRIPTION:
This study would improve the localization of the epileptogenic zone and reduce the overall duration of monitoring, especially in patients who do not experience a sufficient number of seizures during the implantation period. In addition, it would be possible to use micro-electrodes and propose a better surgical treatment to some patients whose preliminary assessment with macro-electrodes has not provided significant results. Finally, the data collected during this study will help us to further understand pathological brain activity and to describe the neuronal circuitry that gives rise to cortical signals and the relationships between them (from spindles to high frequency oscillations).

ELIGIBILITY:
Inclusion Criteria:

* inclusion criteria is determined based on the clinical diagnosis of the refractory epilepsy and the admissibility of the patient for the stereoelectroencephalography (sEEG) procedure

Exclusion Criteria:

* severe psychiatric disorders,
* severe agitation during their crisis
* contraindication for performing an MRI: claustrophobia, a cardiac or neural stimulator, ferromagnetic surgical clips, cochlear implants, intraocular metallic foreign body or in the nervous system,
* contraindication to intracerebral investigation (macro-electrodes): ongoing infection, severe associated pathology (cardiac, pulmonary, renal, hepatic), pregnant or nursing women,
* anti thrombotic ongoing treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
evaluate the recording of fast ripples (FRs) and single neuron activity in the brain with the micro tetrodes | 1 week after implant
  sum of number of single units recorded and the number of fast ripples (FRs)

SECONDARY OUTCOMES:
Efficiency of microelectrodes compared to macroelectrodes | 10 days after implant
  proportion and quality of the FRs recorded by the macro-blocks immediately adjacent to the microelectrodes located in the EZ

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided